CLINICAL TRIAL: NCT07085403
Title: Let's CO-OPerate! Together we Are Stronger: Exploring the Effectiveness of the CO-OP Cognitive Problem-solving Approach in the Context of an Intensive Group Rehabilitation Training for a Paediatric Population With Executive Function Deficits and/or Developmental Coordination Disorders Following Brain Injury
Brief Title: Let's CO-OPerate! Together we Are Stronger
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Principal Investigator, Hélène LEBRAULT, principal investigator, Hopitaux de Saint-Maurice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COOPerons - PR- 2024 - 7
Record Dates: First submitted 2025-07-04; First posted 2025-07-25 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Executive Function Deficits (EFD); Developmental Coordination Disorder; Acquired Brain Injury (Including Stroke); Brain Injury, Fetus and Neonate
Keywords: paediatric rehabilitation; occupational therapy; executive function deficits; developmental coordination disorder; acquired brain injury; fetus and neonate brain injury; Cognitive Orientation to daily Occupational Performance (CO--OP); intensive training; individual and group rehabilitation
MeSH Terms: conditions — Motor Skills Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: replicated single case experimental study using a randomized multiple baseline design across participants and goals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COOP experimental arm (Experimental)
  Interventions: Other: Cognitive Orientation to daily Occupational Performance (CO-OP) is a cognitive problem-solving approach

INTERVENTIONS:
Other: Cognitive Orientation to daily Occupational Performance (CO-OP) is a cognitive problem-solving approach — Cognitive Orientation to daily Occupational Performance (CO-OP; CO-OP approach) is a performance-based treatment approach for children and adults who experience difficulties performing the skills they want to, need, to or are expected to perform. CO-OP is a specifically tailored, active client-centered approach that engages the individual at the meta-cognitive level to solve performance problems. Focused on enabling success, the CO-OP approach employs collaborative goal setting, dynamic performance analysis, cognitive strategy use, guided discovery, and enabling principles. These elements, all considered essential to the CO-OP Approach, are situated within a structured intervention format, and may involve the parent/significant other as appropriate.

SUMMARY:
The goal of this replicated single case experimental study using a randomized multiple baseline design across participants and goals is to enable children/adolescents (aged 8-16 years) with developmental coordination disorders and/or executive function deficits following an acquired or congenital brain injury, to achieve their occupational goals. The aim is to make them more independents and autonomous in their daily lives. To achieve this, we're going to offer them an intensive group CO-OP (Cognitive Orientation to daily Occupational Performance Approach) rehabilitation training, and actively involving the parents. The main questions it aims to answer are:

* To evaluate the improvement in occupational performance* (and its maintenance over time) following intervention using the CO-OP Approach.

  *Occupational performance is a person's ability to choose, organize and engage in meaningful occupations that give them satisfaction. These occupations, determined by culture and corresponding to their age group, enable them to take care of themselves, have fun and contribute to the social and economic fabric of the community.
* To gather parents' experiences of supporting their child during the CO-OP intervention and its follow-up phase.

Participants will be asked to identify 3 goals that they would like to achieve with the CO-OP Approach. The CO-OP intervention will take the form of two half-days a week for 5 weeks, with 1 hour 30 minutes of individual CO-OP sessions and 1 hour 30 minutes of group sessions.

ELIGIBILITY:
Inclusion criteria:

* Children/adolescents (8-16 years old) with coordination disorders and/or executive function deficits, following a acquired brain injury more than 3 months ago or a congenital brain lesion or a neurodevelopmental disorder.
* Executive function deficits as assessed by neuropsychological tests (standardised tests and/or questionnaires) and/or coordination disorders as assessed by neuropsychological tests (standardised tests and/or questionnaires).
* Vision and hearing normal or sufficient to communicate effectively (with appropriate correction where necessary).
* Cognitive, behavioural and expressive/receptive communication skills enabling them to identify goals and participate actively in the CO-OP intervention process.
* Membership of a health insurance scheme or beneficiary.
* Agreement of the child/adolescent and informed consent expressed by at least one of the holders of parental authority.

Non-inclusion criteria :

* Children/adolescents who do not meet the inclusion criteria.
* Children/adolescents and/or parents non-French-speaking.
* Presenting intellectual difficulties, or severe problems of comprehension, memory or attention, as described in the CO-OP recommendations.
* A diagnosed severe anxiety-depressive disorder that is not compatible with participation in the study.
* Inability to remain involved until the end of the CO-OP intervention phase (e.g. planned move).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale (GAS) | Baseline to 6-months post-intervention: two times per week during baseline and intervention phase for each chosen-goal ; one time at 2, 4 and 6-months post-intervention.
  The Goal Attainment Scale (GAS) is a criterion--referenced measure used to quantify the degree to which personal goals are achieved. GAS methodology consists in:
  * Defining a rehabilitation goal;
  * Choosing an observable behaviour that reflects the degree of goal attainment;
  * Defining the patient's initial level with respect to the goal;
  * Ranging from a ''no change'' to a ''much better than expected outcome'');
  * Evaluating the patient after a defined time interval;
  * Calculating the overall attainment score for all the rehabilitation goals. A five-point scale will be used: "-2" is the initial pretreatment level; "-1" represents progression towards the goal without goal attainment; ''0'' is the expected level after treatment, (and therefore, the ''most likely'' level after treatment); ''+1'' represents a better outcome than expected; ''+2'' is the best possible outcome that could have been expected for this goal.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Once before baseline, at immediate post-intervention, at 2, 4 and 6-months post-intervention.
  The Canadian Occupational Performance Measure is an individualized, client--centered, semi--structured interview used to identify occupational performance issues.For each performance issue, perceived performance and satisfaction are scored on a 1 to 10 Likert scale.
  Performance and satisfaction are rated by children and parents on a scale of 1 to 10 (1= not at all able to perform the activity (performance) / not at all satisfied with the way the activity is performed (satisfaction); 10 = perfectly able to perform the activity (performance) / perfectly satisfied with the way the activity is performed (satisfaction). A difference of 2 points between pre- and post-intervention is clinically significant.
  For each self--identified goal, four different COPM ratings will be obtained: (1) the participant's perceived occupational performance rating; (2) the participant's satisfaction rating; (3) the parent's perceived occupational performance rating; (4) the parent's satisfaction rating.
Behavior Rating Inventory of Executive Function questionnaire (BRIEF) | twice in baseline, once in immediate post-intervention and once at 2,4,6 month post-intervention.
  The Behavior Rating Inventory of Executive Function questionnaire (BRIEF, or BRIEF-A for adults'version) provide an ecological assessment of executive functioning through its repercussions in family and school context. Currently, this questionnaire is the best validated and most widely used in children in various congenital, developmental or acquired conditions. The outcome measure is the Global Executive Composite score (GEC) T-Scores (Mean: 50; SD: 10; clinical range cutoff: T-Scores≥65).
Entretien Engagement des Proches | once at immediate post-intervention, 4 and 6 months-post-intervention]
  The aim of this interview is to collect information on the experience of use of CO-OP by family caregivers with the participant, outside of rehabilitation sessions. No scale of score, the interviews will be analyzed according to a qualitative description.

OTHER OUTCOMES:
Behavioural Assessment of the Dysexecutive Syndrome for Children (BADS-C) (aged 8-- 15 years) | Once before the baseline for children aged 8-15 years
  Behavioural Assessment of the Dysexecutive Syndrome for Children (BADS-C) predicts everyday problems associated with a major area of cognitive deficit that can impede functional recovery and the ability to respond to rehabilitation programs. The therapist can be use 2 subtests to assess the executive functions deficits (Zoo Part 1 and 2 subtest; Six parts subtest). Standard scores: mean 10 (SD: 3).
Behavioural Assessment of the Dysexecutive Syndrome (BADS) (participants aged 16 years) | Once before the baseline for participants aged 16 years
  Behavioural Assessment of the Dysexecutive Syndrome (BADS) predicts everyday problems associated with a major area of cognitive deficit that can impede functional recovery and the ability to respond to rehabilitation programs. The therapist can be use 2 subtests to assess the executive functions deficits (Zoo Part 1 and 2 subtest; Six elements subtest). Standard scores : means 10 (SD: 3).
Movement Assessment Battery for Children (M-ABC) | once before the baseline
  The M-ABC is designed to identify and describe impairments in motor performance of children and adolescents. It will be use to assess developmental coordination disorders. Standard scores: mean 10 (3).
Wechsler Intelligence Scale for Children (WISC) | once before the baseline
  Wechsler Intelligence Scale for Children is an intelligence test that measures a child's intellectual ability and 5 cognitive domains that impact performance. This test (or equivalent, depending on the neuropsychologist's decision) will be used to assess development coordination disorders and/or executive function deficits. Standard scores for index: mean 100 (SD: 15); Standard scores for subtests: mean 10 (SD: 3).
Children Cooking Test (CCT) | once before the baseline
  The Children's Cooking Task (CCT) is a complex test that has been specifically developed to assess executive functions in a standardized open-ended environment (cooking). The CCT can be used by therapists to assess executive function deficits. Number of errors / z score (compared to age-matched controls); Task duration (min) / z score (compared to age-matched controls).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Paris-Est Val-de-Marne, Saint-Maurice, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steenbeek D, Ketelaar M, Galama K, Gorter JW. Goal Attainment Scaling in paediatric rehabilitation: a report on the clinical training of an interdisciplinary team. Child Care Health Dev. 2008 Jul;34(4):521-9. doi: 10.1111/j.1365-2214.2008.00841.x. PMID 19154553
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506